CLINICAL TRIAL: NCT02425358
Title: Timing for Intracoronary Administration of Bone Marrow Mononuclear Cells After Acute ST-elevated Myocardial Infarction: a Pilot Study
Brief Title: Timing for Bone Marrow Mononuclear Cells After Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Rchuang, Professor, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004BA714B05-2
Record Dates: First submitted 2015-04-15; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Myocardial Infarction
Keywords: cell therapy; BMC; timing
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMC therapy within 24 hours (Experimental): Patients with acute myocardial infarction who receive intracoronary infusion of BMC within 24 hours after successful primary PCI.
  Interventions: Other: BMC therapy within 24 hours
- BMC therapy within 3-7 days (Experimental): Patients with acute myocardial infarction who receive intracoronary infusion of BMC within 3-7days after successful primary PCI.
  Interventions: Other: BMC therapy within 3-7 days
- BMC therapy within 7-30 days (Experimental): Patients with acute myocardial infarction who receive intracoronary infusion of BMC within 7-30days after successful primary PCI.
  Interventions: Other: BMC therapy within 7-30 days
- PCI only (Active Comparator): Patients with acute myocardial infarction who were performed successful primary PCI.
  Interventions: Other: PCI only

INTERVENTIONS:
Other: BMC therapy within 24 hours — The BMCs were isolated by Ficoll density gradient centrifugation on Lymphocyte Separation Medium. BMCs were infused into IRA at the site of the previous occlusion. This was accomplished with the use of a microtubular. After positioning of the microtubular into the distal segment vessel of the stent position in the infarct-related artery, 15 milliliter of the whole cell suspension was slowly administered via microtubular. The usual time should be over 10min to prevent back-flow and to prolong cellular contact time for cellular migration into the tissue. Patients in BMC therapy group within 24 hours remained in the cath-lab until the entire procedure, including primary PCI and intracoronary BMC infusion, was completed.
  Arms: BMC therapy within 24 hours
Other: BMC therapy within 3-7 days — Patients in this group, who underwent a second procedure, to receive BMC transplantation in the cath-lab during the same hospitalization or returned for a second hospitalization.
  Arms: BMC therapy within 3-7 days
Other: BMC therapy within 7-30 days — Patients in this group, who underwent a second procedure, to receive BMC transplantation in the cath-lab during the same hospitalization or returned for a second hospitalization.
  Arms: BMC therapy within 7-30 days
Other: PCI only — The saline was intracoronary infusion with the use of microtubular.
  Arms: PCI only

SUMMARY:
Most studies on intracoronary bone marrow mononuclear cell (BMC) transplantation for acute myocardial infarction (AMI) involve treatment 3-7 days after primary percutaneous coronary intervention (PCI); however, the optimal timing is unknown. The present study assessed the therapeutic effect at different times after ST-elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
On the basis of experimental studies that bone marrow mononuclear cells (BMCs) transfer in the injured tissue can promote regional myocardial perfusion and improved cardiac function, several clinical trials have shown that intracoronary bone marrow mononuclear cell (BMC) transplantation in acute myocardial infarction (AMI) patients several days after myocardial reperfusion is safe and may enhance the improvement of left ventricular ejection fraction (LVEF). The timing of BMC administration, baseline LVEF, dosage of BMC and other factors has been linked to improvement in LVEF after BMC transplantation. In our previous work, we gave BMCs within 24 hours after emergency percutaneous coronary intervention (PCI) and found that it was safe and effective . In addition, there are another report about longer time from symptom onset to BMC infusion (2-4 weeks), which also appeared effective . The timing of intracoronary stem cell administration may have a critical effect on cell engraftment and may be responsible for the various biological and functional responses to therapy. However, few studies have directly addressed the optimal timing of cell injections. Therefore, in this prospective randomized study, BMCs were given at different times (within 24 hours, 3 to 7 days, or 7 to 30 days after reperfusion) to investigate whether the timing of therapy affects the therapeutic response of AMI patients.

ELIGIBILITY:
Inclusion Criteria:

* a history of first acute ST-elevation myocardial infarction
* treatment with successful PCI two to twelve hours after symptom onset
* LVEF less than 50% on angiography immediately after emergency PCI or rescue PCI

Exclusion Criteria:

* previous Q-wave myocardial infarction
* cardiogenic shock
* severe coexisting conditions such as acute and chronic heart failure, malignant
* arrhythmia, renal failure and severe bleeding that interfered with the ability of the
* patient to comply with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change of left ventricular eject factor (LVEF) from the baseline | 12 months

SECONDARY OUTCOMES:
Change of left ventricular end-diastolic volume (LVESV) from the baseline | 12 months
Change of left ventricular end-systolic volume (LVEDV) from the baseline | 12 months
Change of myocardial perfusion from the baseline | 12 months

REFERENCES:
- [Background] Yao K, Huang R, Sun A, Qian J, Liu X, Ge L, Zhang Y, Zhang S, Niu Y, Wang Q, Zou Y, Ge J. Repeated autologous bone marrow mononuclear cell therapy in patients with large myocardial infarction. Eur J Heart Fail. 2009 Jul;11(7):691-8. doi: 10.1093/eurjhf/hfp062. Epub 2009 May 6. PMID 19420003
- [Background] Yao K, Huang R, Qian J, Cui J, Ge L, Li Y, Zhang F, Shi H, Huang D, Zhang S, Sun A, Zou Y, Ge J. Administration of intracoronary bone marrow mononuclear cells on chronic myocardial infarction improves diastolic function. Heart. 2008 Sep;94(9):1147-53. doi: 10.1136/hrt.2007.137919. Epub 2008 Apr 1. PMID 18381377
- [Derived] Huang R, Yao K, Sun A, Qian J, Ge L, Zhang Y, Niu Y, Wang K, Zou Y, Ge J. Timing for intracoronary administration of bone marrow mononuclear cells after acute ST-elevation myocardial infarction: a pilot study. Stem Cell Res Ther. 2015 May 29;6(1):112. doi: 10.1186/s13287-015-0102-5. PMID 26021558